CLINICAL TRIAL: NCT05031533
Title: A Prospective Study on the Efficacy, Safety and Immune Effects of Dose-painting Radiation for Locally Advanced Non-small Cell Lung Cancer(LA-NSCLC)
Brief Title: Dose-painting Radiation for LA-NSCLC
Acronym: DPRLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, LI TAO, Researcher, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCHEC202108
Record Dates: First submitted 2021-08-25; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Non-small Cell Lung Cancer Stage III; Non-small Cell Lung Cancer Stage II
Keywords: radiotherapy; dose-painting radiation; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Radiation therapy: Dose-painting radiation
  Systemic treatment: Choose a systemic treatment plan according to the patient's genetic testing status
  (1) Chemotherapy
  1. Squamous cell carcinoma: Paclitaxel 135mg/m2 D1 + Cisplatin 25mg/m2 D1-3, every 21 days, a total of 2-4 cycles.
  2. Non-squamous cell carcinoma (adenocarcinoma, large cell carcinoma): Pemetrexed 500mg/m2 d1 + Cisplatin 75 mg/m2 d1-3, a total of 2-4 cycles.
  (2) Targeted therapy: According to the patient's genetic testing status, molecular targeted therapy such as EGFR-TKI and ALK inhibitors can be selected; (3) Immunotherapy: According to the patient's genetic testing status, immunotherapy such as PD1/PD-L1 inhibitors can be selected;
  Interventions: Radiation: Dose-Painting Radiation

INTERVENTIONS:
Radiation: Dose-Painting Radiation — Radiation therapy:
  1. Delineation of target area:
     The primary tumor is delineated into different target areas according to the anatomical position of the tumor, including the central area tumor GTV-Tcentral and GTV-Tperipheral.
  2. Exposure dose:
  1) GTV-Tcentral: 2.0～2.5Gy/f, bid, 10-13d, physical dose 40-65Gy 2) GTV-Tperipheral: 3.0～4.0Gy/f, bid, 10-13d, physical dose 60-104Gy 3) GTV-N (mediastinal lymph node): 2.0Gy/f, bid, 10-13d, physical dose 40-52Gy

SUMMARY:
The study evaluated the effectiveness, safety and immune effects of dose-painting radiation in patients with locally advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
The study evaluated the effectiveness, safety and immune effects of dose-painting radiation in patients with locally advanced non-small cell lung cancer.

The primary endpoint is PFS. Secondary points contains ORR, OS, HRQoL, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or the legal representative of the patient can sign a written informed consent, and can understand and agree to follow the research requirements;
2. The age at the time of signing the informed consent form is between 18 and 75 years old;
3. It is diagnosed as non-small cell lung cancer by histology, and is suitable for radical radiotherapy:
4. Stage II-Ⅲ (AJCC 8th edition [Rice et al., 2017]) inoperable NSCLC patients (not medically suitable for surgery or refuse surgical intervention);
5. Measurable lesions that meet the definition of RECISTv1.1;
6. ECOG physical status ≤ 2;
7. Survival expectancy ≥ 3 months;
8. Hemoglobin ≥100g/L, WBC≥4×109/L, platelet ≥100×109/L (or follow the standards of each center);
9. Liver function: ALT, AST<1.5 times the upper limit of normal (ULN), total bilirubin<1.5×ULN;
10. Renal function: serum creatinine <1.5×ULN;
11. Pulmonary function: FEV1>50%, the percentage of DLCO (lung diffusion function) measured value and predicted value>80% mild to moderate lung function impairment.
12. The patient has good compliance with the treatment and follow-up.

Exclusion Criteria:

1. There is evidence of distant metastasis (M1, AJCC 8th edition [Rice et al., 2017]);
2. There is pleural effusion, pericardial effusion or ascites that is not clinically controlled and requires repeated drainage or medical intervention (within 2 weeks before randomization);
3. Intolerance or resistance to the chemotherapy, targeted, and immunotherapy specified in the experimental protocol;
4. Have received radiotherapy and surgical treatment;
5. There were other active malignant tumors ≤ 2 years before enrollment, except for the specific cancers under study in this study and locally recurring cancers that have been cured (eg, resected basal cell or squamous cell skin cancer, superficial Bladder cancer, carcinoma in situ of the cervix or breast);
6. A history of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases, including pulmonary fibrosis, acute lung diseases, etc.;
7. Has suffered from other malignant tumors;
8. Subjects who have received other drug trials within the past month;
9. Pregnant or lactating women and women who refuse contraception during the treatment observation period;
10. People with a history of severe allergies or idiosyncratic physique;
11. Those with a history of severe lung or heart disease;
12. Refusal or inability to sign the informed consent to participate in the trial;
13. Drug or alcohol addicts;
14. Personality or mental illness, lack of capacity for civil conduct or limited capacity for civil conduct.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
FPS | up to 3 years
  progression-free survival (PFS) refers to the time from enrollment to the first recording of disease progression as determined by RECISTv1.1, or to death due to any cause (whichever occurs first). PFS will be analyzed in the ITT analysis set.

SECONDARY OUTCOMES:
ORR | up to 3 years
  Objective response rate, according to RECISTv1.1, the proportion of patients with CR or PR was determined. If the patient has not undergone a post-baseline assessment, it is considered unremission
OS | up to 3 years
  OS(Overall survival) refers to the time from enrollment to the first recorded death due to any cause (whichever occurs first).
HRQoL | up to 3 years
  HRQoL uses EORTCQLQ-C30 to assess the overall health of patients. The post-baseline score of the treatment group was studied, and the score changes from the baseline were summarized descriptively.

OTHER OUTCOMES:
Prognostic Biomarkers | up to 8 weeks
  The expression of lymphocyte subsets in peripheral blood, including CD3+ T cells, CD4+ T cells, CD8+ T cells, CD8+CD28+ T cells, CD8+CD28- T cells, Treg cells, NK cells, NKT cells, γδ T cells;
Prognostic Biomarkers | up to 8 weeks
  The changing trend of various cytokines in radiotherapy, including IL-6, IL-1b, IL-9, TNF-a, TGF-β, IL-10, IL-21, etc.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sichuan Cancer Hospital & Institute, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming
  - Chongqing university three Gorges hospital, Wanzhou
  - General Hospital of Ningxia Medical University, Yingchuan

IPD SHARING:
Plan to Share IPD: Undecided